CLINICAL TRIAL: NCT03454308
Title: Patient Centered Health Technology Medication Adherence Program for African American Hypertensives
Acronym: SMASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 452; HL130917 (Other: NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-03-05 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hypertension; Medication Non-Adherence
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMASH (Experimental): Automated reminder functions activated on pill monitoring device, motivational text messages, at home BP monitoring
  Interventions: Behavioral: SMASH
- Enhanced SC (Other): No reminder functions on the pill monitoring device, attention control text messages
  Interventions: Behavioral: Enhanced SC

INTERVENTIONS:
Behavioral: SMASH — Auditory and visual reminders are active on Pill device will alert subject each time their medication dose is due. Pill device will transmit dose taken time stamps to researchers. Text message the following morning with tailored motivational messages that reflect the medication dose adherence from the preceding day. Subjects will monitor their BP at home at least every third day using Bluetooth monitor linked to smartphone to transmit encrypted readings to researchers.
  Arms: SMASH
Behavioral: Enhanced SC — Auditory and visual reminders are inactive on Pill device. Pill device will transmit dose taken times to researchers. Healthy lifestyle test messages as attention control.
  Arms: Enhanced SC

SUMMARY:
This will be a two--arm Randomized controlled trial (RCT) design that will assess efficacy of the Smartphone Medication Adherence Stops Hypertension (SMASH) mobile health ( mHealth) program compared to an enhanced standard care (SC) program. Participants will be African-American (AA) hypertension patients with no other known chronic diseases.

Participants found to have uncontrolled hypertension (HTN) and medication non-adherence via electronic device monitoring will be randomized to SMASH or enhanced Standard Care (SC). The SMASH group will receive reminders in the form of auditory and visual reminders from a pill monitoring device when their medication dose is due, they will monitor their blood pressure at home and will receive tailored motivational text messages based upon levels of adherence . Enhanced SC group will use the pill monitoring device without reminder functions enabled and will receive text messages on topics of healthy lifestyles not related to medication adherence and hypertension.

The active intervention will continue for 6 months and follow-up will continue for 1 year.

DETAILED DESCRIPTION:
192 AAs (21-59 yrs ) with uncontrolled HTN (no other comorbidities) and Medication Non-Adherence (MNA) will be recruited according to the inclusion and exclusion criteria found elsewhere. In the first phase of screening,resting BP protocols will be performed to determine hypertension is uncontrolled. Only subjects with verified uncontrolled HTN will proceed to the second screening phase .This is a 4 week medication monitoring phase using an electronic medication device with reminder alerts deactivated.Medication non-adherence (MNA) will be determined through medication possession ratio and by the timestamped intake adherence to their predesignated intake schedule across the 4 week period. MA score <0.85 over the 4-week screening and whose subsequent resting BP evaluations reconfirm uncontrolled HTN will be eligible for enrollment into the RCT.

SMASH subjects will have their pill monitor reminder functions activated, start receiving personalized motivational text messages and provided and instructed on use of a validated Bluetooth--enabled BP monitor used at home during the intervention period.

Enhanced SC subjects will continue to use the pill device with reminder functions disabled for another 6 months. In order to control for attention exposure SC subjects will be sent text messages on topics related to healthy lifestyle behaviors (diet, physical activity,no smoke exposure) but not related to Medication Adherence (MA) or HTN.

All subjects will complete 5 study visits where BP,medication possession ratios, and surveys will be completed. 24-hour Ambulatory Blood Pressure (ABP) monitoring will be performed every 6-months (4 times) during the study.

ELIGIBILITY:
Inclusion Criteria:

1. African American or Black, 21--59 years old
2. Prescribed medication(s) only for HTN
3. Medication possession ratio (MPR) <.85 for last 3 months
4. uncontrolled HTN (SBP ≥130 mmHg) based upon last clinic visit within previous 12 months, initial clinic screening & subsequent baseline recruitment evaluation following one month med intake screening with score of <.85
5. 24--hour SBP ≥ 130 mmHg on clinic screening and subsequent recruitment evaluation
6. Ability to speak, hear and understand English
7. Able to take their own BP and self--administer medications
8. Owns smart phone with data plan
9. Primary care provider's assent that patient is able to participate

Exclusion Criteria:

1. No other known chronic disease (e.g., chronic kidney disease (GFR<50 mL/1.7 m2/min;; diabetes (type one or two) renal dialysis cancer diagnosis or treatment in past 2 years prior cv event such as heart attack, congestive heart failure, arterial stent, coronary artery bypass graft psychiatric illness
2. Beck Depression Inventory score >13
3. Ongoing substance abuse (e.g., >21 drinks/week)
4. Planned pregnancy
5. Vulnerable populations such as pregnant or nursing women, prisoners, and institutionalized individuals.

Ages: 21 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Chandler, PhD, Principal Investigator — MUSC College of Nursing
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We will use 8 practice sites in each arm RCT design with clinic as unit of randomization and patient as unit of analysis.
Units Other Than Participants: clinical site
Groups:
- SMASH: Automated reminder functions activated on pill monitoring device, motivational text messages, at home BP monitoring
  SMASH Arm: Auditory and visual reminders are active on Pill device will alert subject each time their medication dose is due. Pill device will transmit dose taken time stamps to researchers. Text message the following morning with tailored motivational messages that reflect the medication dose adherence from the preceding day. Subjects will monitor their BP at home at least every third day using Bluetooth monitor linked to smartphone to transmit encrypted readings to researchers.
- Enhanced SC: No reminder functions on the pill monitoring device, attention control text messages
  Enhanced SC Arm: Auditory and visual reminders are inactive on Pill device. Pill device will transmit dose taken times to researchers. Healthy lifestyle test messages as attention control.
Period: Overall Study
Arm/Group | SMASH | Enhanced SC
Started | 97; 4 clinical site | 107; 4 clinical site
Completed | 97; 4 clinical site | 107; 4 clinical site
Not Completed | 0; 0 clinical site | 0; 0 clinical site

BASELINE CHARACTERISTICS:
Population: Participants were African American Adults with a sole diagnosis of uncontrolled hypertension
Groups:
- Total: Total of all reporting groups
Arm/Group | SMASH | Enhanced SC | Total
Number analyzed (Participants) | 97 | 107 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 107 | 204
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.3) | 47.0 (9.7) | 48.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 74 | 139
  Male | 32 | 33 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 97 | 107 | 204
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 97 | 107 | 204
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 97 | 107 | 204

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Meeting JNC8 Guidelines for BP Control
Description: Percent of subjects meeting JNC8 Guidelines for BP control (<140/90)
Time Frame: at 6 months at the end of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | SMASH | Enhanced SC
Number analyzed (Participants) | 97 | 106
Participants | 97 | 106

2. Primary Outcome: Percent of Participants* With Medication Adherence to >.90" as Accurate and Appropriate
Description: Medication adherence >.90 using electronic medication intake devices. An algorithm is used which takes into account timing of dosage intakes using timestamped data from the devices.
Time Frame: Average across 6 mos.of intervention
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Enhanced SC | SMASH
Number analyzed (Participants) | 40 | 40
percentage of participants | 27.5 (29.4) | 80.3 (9.5)

3. Secondary Outcome: Changes in Medication Adherence Self-Efficacy
Description: Changes in Medication Adherence Self-Efficacy (MASES-R) with increased self-efficacy (higher scores) desired. (attached) (Range: 1-4)
Time Frame: Months 1 and 6
Reporting Status: Not Posted

4. Secondary Outcome: Percent Achieving and Sustaining 24-hr BP Control (< 130/80 mmHg)
Description: 24-hr ABP BP average SBP to (< 130/80 mmHg) - 0 participants with this data reported. Our technology team changed half way through the trial and our ability to use the 24 hour ambulatory monitors code that was built within our institution and transfer it to use with the external data team was unsuccessful.
Time Frame: Month 6 of intervention period and at month 6 and 12 of follow-up period.
Reporting Status: Not Posted, anticipated posting 2050-01

5. Secondary Outcome: Changes in Autonomous Motivation
Description: Changes in Autonomous Motivation Questionnaire with increase in Relative Autonomy Index desired. (Attached)(Range -36 to 36)
Time Frame: Months 3,6 of intervention period and at months 6 and 12 of follow-up period.
Reporting Status: Not Posted

6. Secondary Outcome: Percent of Subject Achieving and Maintaining JNC8 Guidelines for BP Control (<140/90)
Description: Percent of subject achieving and maintaining JNC8 Guidelines for BP control (<140/90)
Time Frame: Month 6 of intervention and months 6 and 12 of follow-up period
Reporting Status: Not Posted

7. Secondary Outcome: Percent of Subjects Achieving and Maintaining Medication Adherence >.90.
Description: Percent of subjects achieving and maintaining Medication Adherence >.90.
Time Frame: Months 3,6 of intervention period and at months 6 and 12 of follow-up period.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 18 months
Arm/Group | SMASH | Enhanced SC
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/107
Other Adverse Events (participants affected / at risk) | 0/97 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03454308/Prot_SAP_001.pdf
  • Informed Consent Form (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03454308/ICF_000.pdf